CLINICAL TRIAL: NCT02508350
Title: The Pharmacokinetics and Pharmacodynamics of High-dose Daptomycin in Patients With Septic Shock
Brief Title: The Pharmacokinetics/Pharmacodynamics of High-dose Daptomycin in Patients With Septic Shock
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhongda Hospital (Other)
Responsible Party: Principal Investigator, Yingzi Huang, Chief Physician, Zhongda Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 2015Dapto
Record Dates: First submitted 2015-07-18; First posted 2015-07-24 (Estimated); Last update posted 2015-07-24 (Estimated); Status verified 2015-07

CONDITIONS: Septic Shock
MeSH Terms: conditions — Shock, Septic | interventions — Daptomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- daptomycin (Experimental): Daptomycin for injection 10-12mg/kg/day,determination of plasma concentration
  Interventions: Drug: Daptomycin; Other: determination of plasma concentration

INTERVENTIONS:
Drug: Daptomycin — Drug: Daptomycin for Injection（Cubicin,AstraZeneca） dosage: 10-12mg/kg/day frequency: once a day duration: 14 days
  Other Names: Cubicin
Other: determination of plasma concentration — A maximum of 12 blood samples (1.5mL) were collected in Ethylenediaminetetraacetic acid disodium salt (EDTA-Na2) tubes over a 6-dose administration sequence.Sampling was done prior to the administration of the first dose, at 30 minutes (end of infusion),and at 4,12,and 24 hours after the initial dose.Additional blood samples were collected at the end of infusion (peak) and prior to the subsequent dose (trough) for doses 2-5.After the sixth dose the blood samples were collected prior to the administration and at 4,and 24 hours after the end of infusion.

SUMMARY:
The first objective of this study was to characterize the pharmacokinetics and pharmacodynamics of daptomycin with a daily dose of 12mg/kg in septic shock patient; the second objective is to identify the optimal dosing scheme for daptomycin among patients with septic shock and to enhance therapeutic outcomes.

DETAILED DESCRIPTION:
Daptomycin is a novel lipopeptide exhibiting concentration-dependent bactericidal activity against multidrug-resistant Gram-positive pathogens, including Methicillin-resistant Staphylococcus aureus (MRSA). In recent years, daptomycin plays an important role in the treatment of septic shock. The pharmacokinetics of daptomycin is significant changed in patients with septic shock, it is proved that the recent dosage regiment comes with a low blood drug concentration and unsatisfactory outcome. Although the high-dose daptomycin shows safety and effectiveness in the treatment of critically ill patient, but still the pharmacokinetics and pharmacodynamics data is scant. So the purposes of this study is to characterize the pharmacokinetics and pharmacodynamics of daptomycin with a daily dose of 12mg/kg in septic shock patient; the second objective is to identify the optimal dosing scheme for daptomycin among patients with septic shock and to enhance therapeutic outcomes.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years and ≤75 years
* confirmed or suspected bloodstream and soft tissue infections caused by a grampositive organism

Exclusion Criteria:

* known hypersensitivity to daptomycin or product excipients
* documented or suspected pneumonia caused by a grampositive organism
* infection with a daptomycin-resistant organism
* presence or history of rhabdomyolysis
* signs or symptoms of myopathy with an elevation of creatine phosphokinase concentrations 6.pregnancy or breast-feeding

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2015-01; Primary Completion 2015-12 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Area under the curve(AUC)/Minimum inhibitory concentration(MIC) | 6 days
Peak concentration (Cmax)/Minimum inhibitory concentration(MIC) | 6 days

SECONDARY OUTCOMES:
mortality rate | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Yingzi - Huang, Study Director — southeast univerity, China
Locations (1):
- Zhongda hospital, Southeast University, Nanjing, Jiangsu, China